CLINICAL TRIAL: NCT01105871
Title: Subjective Analgesic Effects of Naloxone and Virtual Reality
Acronym: Narcan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Sam Sharar, Principal Investigator, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 35974-D
Record Dates: First submitted 2010-03-19; First posted 2010-04-19 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Pain
Keywords: Pain relief
MeSH Terms: conditions — Pain | interventions — Naloxone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- naloxone (Active Comparator): 4 mg in 10 ml saline iv bolus
  Interventions: Drug: naloxone
- saline placebo (Placebo Comparator): 10 ml of normal saline iv bolus
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: naloxone — 4 mg naloxone in 10 ml saline given iv bolus
  Other Names: Naloxone = Narcan
  Arms: naloxone
Drug: Placebo — 10 ml of normal saline iv bolus
  Arms: saline placebo

SUMMARY:
This study is designed to test a specific hypothesis exploring the neurophysiologic mechanism(s) that underlie the pain- relieving effects of immersive Virtual Reality (VR) as a non-pharmacologic pain management technique, using healthy volunteers experiencing carefully controlled thermal and/or electrical pain in the laboratory. Over the past decade, our research group has performed a series of NIH-funded investigations of VR analgesia - in both the clinical pain and laboratory pain settings - demonstrating its clinical efficacy and safety. In the current study we will test pharmacologic manipulation of VR analgesia (with the opioid analgesia antagonist naloxone). We anticipate that this theoretical work will provide a foundation for future clinical applications of immersive VR - whether used alone or in combination with other analgesic agents - and make immersive VR a more effective and more widely used analgesic tool for the treatment of clinical pain.

Our previous work with immersive VR indicates that its use during a painful event can reduce subjective pain reports during both acute clinical and laboratory pain by 20-50% [1]. Furthermore, we have shown that effective VR analgesia is associated with reduced pain-related brain activity that is quantitatively and qualitatively comparable to clinically relevant doses of systemic opioid analgesics [2]. The laboratory pain protocol proposed in the current application is identical to the UW HSD-approved protocol used in our previous studies (#25296 - "Reducing Brief Thermal and Electrical Pain"). What is specifically different in the current protocol is the use of naloxone to determine whether VR analgesia operates through an endogenous opioid-dependent mechanism or not. The results of this study will not only suggest the mechanism of action of VR analgesia, but also allow us to more effectively apply immersive VR analgesia in the clinically pain setting through its thoughtful combination with well-established pharmacologic analgesic techniques, such as opioid analgesia administration.

The specific aim of this study and the hypothesis it tests are as follows: To determine the extent to which subjective analgesic effects of VR analgesia are inhibited by opioid receptor antagonism with naloxone. Hypothesis - VR analgesia will not be inhibited by systemic opioid receptor antagonism, suggesting that VR analgesia is not mediated by release of endogenous opiates and/or by activation of opioid-dependent descending central nervous system pathways.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between the ages of 18 and 60 years
* Ability to communicate orally
* Body mass index of 30 or less

Exclusion Criteria:

* Women who are pregnant, trying to become pregnant or who are breastfeeding.
* History of alcohol or substance abuse
* Major medical illness, including history or migraine headaches
* Allergy or sensitivity to narcotics or naloxone
* Current use of analgesics including acetaminophen, non-steroidal anti-inflammatories, or opioids
* Predisposition to severe motion sickness
* Unusual sensitivity or lack of sensitivity to pain
* Sensitive skin
* Urine toxicology positive for opioids

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-08; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Pain scoring from sessions where naloxone is given or placebo.Pain scoring is a questionnaire using analog scale (1-10). | Outcome measurements will be assessed when all research and analysis has been completed. We project the approximate time frame to be about 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel R Sharar, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States